CLINICAL TRIAL: NCT05387629
Title: The Effect of Social Media in Improving the Academic Achievement of Nursing Students: A Randomized Controlled Study
Brief Title: The Effect of Social Media in Improving the Academic Achievement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Bahar Ciftci, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 80131151/2000302016
Record Dates: First submitted 2022-05-19; First posted 2022-05-24 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Nursing Caries
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Social media increases the academic success of nursing students.
  Interventions: Behavioral: Education
- Control (No Intervention): Social media does not affect the academic success of nursing students.

INTERVENTIONS:
Behavioral: Education — Nursing students will be trained through social media.
  Arms: Experimental

SUMMARY:
In today's living conditions, technology is present in every aspect of our lives and is constantly changing and developing. Thanks to technological developments, progress has been made in the field of communication as well as in many other fields, and this has provided the opportunity to access information quickly. Especially the widespread use of mobile phones has facilitated communication. Thanks to smartphones, which are an integral part of daily life, we can quickly access or share information. Especially with smart phones, interactive access is provided through Social Media, which is one of the most advanced communication tools of our age. Commonly used social media tools are Social Networking websites (Facebook, Twitter, Instagram) in our country and around the world. Social media tools have many features for the development of educational processes. Social media can be used in educational processes to improve communication skills of students and teachers, expand participation, strengthen peer support, and realize cooperative learning. Social media teaching processes; It also provides opportunities such as supporting the learning process of students by enriching it with materials such as pictures, text, video, audio, and supporting the teacher's teaching and evaluation process.

The purpose of this research; To evaluate the effect of social media in improving the academic success of nursing students.

DETAILED DESCRIPTION:
The population of the research will be Atatürk University Nursing Faculty 2nd year students. The sample will consist of students who meet the research criteria, accept the research and use Instagram as social media.

Prior to the study, a priori power analysis was performed to determine the sample size in this study. In the power analysis, it was determined that the sample size should be 80, 40 interventional and 40 control, at a significance level of 0.05, with a confidence interval of 95%, for power of 95% and with a margin of error of 5%.

Inclusion criteria for the study

* Those who agreed to participate in the research
* Students using Instagram
* Those who have a smart mobile phone
* Those who do not have internet problems
* Those who are not absent throughout the research. Exclusion criteria for research
* 2nd year nursing students who did not accept to participate in the research
* Students who do not use Instagram

  * Data collection tools:

"Personal Information Form", "Achievement Test 1" and "Achievement Test 2" will be used in data collection. In addition, psychomotor "Skill Checklists" will be used with OSCE.

Personal Information Form: The questionnaire contains questions such as age, gender, marital status, family structure, and place of residence.

"Achievement Test 1": Multiple choice questions will be prepared by the researchers by scanning the literature. 25 of 50 multiple-choice questions, which are thought to be suitable for the purpose of the research, will be reproduced as the number of students for "Achievement Test 1" and will be kept ready before the application.

The questions in "Achievement Test 1" and "Achievement Test 2" related to the subject of "Parenteral drug applications" will be formed differently from each other.

All students will be taken to the same auditorium at the same time and "Achievement Test 1" will be applied. Evaluation of achievement tests will be made out of 100 points. For this purpose, the total success points of the students will be calculated as 4 times the number of correct answers. The results of "Achievement Test 1" and "Achievement Test 2" will be evaluated with "4" points for each correct answer and "0" points for each wrong answer. The highest score that students can get from achievement tests is "100" and the lowest score is "0".

"Achievement Test 2": Multiple choice questions will be prepared by the researchers by scanning the literature. The remaining 25 questions out of 50 multiple-choice questions prepared previously and 25 of which will be used in "Achievement Test 1" will be arranged for "Achievement Test 2", multiplied by the number of students, and will be kept ready before the application.

The questions in "Achievement Test 1" and "Achievement Test 2" related to the subject of "Parenteral drug applications" will be formed differently from each other. 2 weeks after "Achievement Test 1", all students will be taken to the auditorium at the same time and "Achievement Test 2" will be applied. Evaluation of achievement tests will be made out of 100 points. For this purpose, the total success points of the students will be calculated as 4 times the number of correct answers. The results of "Achievement Test 1" and "Achievement Test 2" will be evaluated with "4" points for each correct answer and "0" points for each wrong answer. The highest score that students can get from achievement tests is "100" and the lowest score is "0".

Skills Checklists: Skills checklists have been developed to be used during clinical skills training and in the objective structured clinical assessment (OSCE) exam to assess students' clinical skill performance. The skill checklists are taken from the "Basic Skills in Nursing Care" book, which shows the application stages of each skill step by step, has been prepared by scanning the relevant current literature, has been used in skill education for 15 years, has been revised at least three times and has undergone editorial review, and published by a national publishing house. There are many basic nursing skills in this book. In the research, parenteral drug administration (IV, ID, SC, IM) checklist will be used to evaluate the skill levels of the students.

*How to collect data: Data will be collected in the Fundamentals of Nursing Course in the fall semester of the 2021-2022 academic year. Nursing Fundamentals Course is one of the compulsory vocational courses in the education of second year nursing students, in which basic nursing skill methods are taught. The course consists of 2 hours of theory and 8 hours of practice. Parenteral drug applications were explained to all students by the same academic staff for 12 hours in the "Basic Care and Clinical Skills Lesson" online due to the pandemic in the spring semester of the 2020-2021 academic year.

In the first stage, an explanation will be given to all students about the research and a "Personal Information Form" will be filled under observation in the classroom environment for students whose consent has been obtained. Afterwards, "Achievement Test 1" will be administered to all students as a pre-test.

Separation of Groups The names of the nursing students who constitute the sample of the research will be written on separate papers and put in a box. From the randomly drawn cards, the first drawn will be in the "interference" group, and the second drawn will be in the "control" group. The process will continue until the papers in the box are exhausted.

In the second stage, a 4-hour theoretical course on the skills aimed to be taught to the students in the intervention and control groups will be explained again. After the theoretical lesson, each skill will be demonstrated in a 2-hour lesson by the instructor in a laboratory environment with the demonstration method in line with the checklists.

In the third stage, videos and informative photos about parenteral drug applications will be shared with the initiative group for 2 weeks from an Instagram page that was created before (@hemsire.notları). This page was created by researchers. After the students in the initiative group are accepted to the page, the privacy setting of the page will be closed and no researcher in the control group will be allowed on the page. Students in the initiative group will be informed that the page's post tracking should be opened. In this way, every shared post will be visible to students. In addition, students in the initiative group will be warned that all posts must be recorded.

In the fourth stage, students in both the intervention and control groups will be applied with task trainer models in the laboratory by taking the checklists as a guide under the supervision of the instructor. Students will practice each skill on the model.

*Evaluation of data: SPPS 23.0 (Statistical Program for Social Sciences) package program will be used to evaluate the data obtained from the research. The conformity of the variables to the normal distribution will be examined using visual (histograms, probability plots) and analytical methods (Kolmogorov-Smirnov test). When comparing control and intervention groups, independent groups t-test will be used for comparisons between normally distributed continuous variables, and chi-square test will be used for categorical variables. If the data from the comparison of the scale scores before and after the application in the intervention group show normal distribution, the paired t test will be applied, and if it does not show normal distribution, the Wilcoxon test will be applied. The relations of the variables with each other will be evaluated by using pearson correlation analysis for normally distributed values and using spearman correlation analysis for non-normally distributed values. Statistical significance level will be accepted as p<0.05.

*Difficulties and limitations of the study: The limitation of this research is that it is carried out only with 2nd year nursing students studying at a university's nursing faculty.

ELIGIBILITY:
Inclusion Criteria:

* Those who agreed to participate in the research
* Students using Instagram
* Those who have a smart mobile phone
* Those who do not have internet problems
* Those who are not absent throughout the research.

Exclusion Criteria:

* 2nd year nursing students who did not accept to participate in the research
* Students who do not use Instagram

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
SOCIAL MEDIA SCALE IN NURSING EDUCATION | 3 months
  Social Media Scale in Nursing Education (HESMÖ): Rodríguez et al. (2021), the scale that determines the use of social media in nursing education consists of 13 items. The scale is in the form of a 5-point Likert (1: strongly disagree-5: strongly agree). The scale consists of 3 sub-dimensions. The first sub-dimension is social media use in nursing education, the second sub-dimension is attitude, and the third sub-dimension is contrast information. High scores obtained from the scale indicate that the level of social media use in nursing education is high. Rodríguez et al. (2021), while the Cronbach's Alpha value was specified as 0.84, the Cronbach's Alpha value was found to be 0.87 in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Bahar Çiftçi, Study Director — Ataturk University
Locations (1):
- Atatürk University Faculty of Nursing, Erzurum, Turkey (Türkiye)